CLINICAL TRIAL: NCT04668274
Title: A Phase 1 Study to Assess the Pharmacokinetics and Safety of Ascending Doses of JOTROL Oral Gelcaps in Healthy Subjects, and to Determine the Influence of Food
Brief Title: JOTROL PK, Safety, and Food Effect Assessment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jupiter Orphan Therapeutics Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol 202016; R44AG067907-01A1 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Results first posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics; Safety; Food-drug Interaction
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) (Experimental): Participants received JOTROL (resveratrol) 200 (2*100) milligram (mg) (Treatment A), gelatin capsule (gelcap), orally, once on Day 1 in fasted conditions in Study Period 1.
  Interventions: Drug: 200 mg resveratrol as JOTROL
- Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) (Experimental): Participants who completed Study Period 1 received JOTROL (resveratrol) 500 (5*100) mg (Treatment B), gelcap, orally, once on Day 1 in fasted conditions in Study Period 2. A 14 days washout period was maintained in study period 1 and 2.
  Interventions: Drug: 500 mg resveratrol as JOTROL
- Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) (Experimental): Participants who completed Study Period 2 received JOTROL (resveratrol) 700 (7*100) mg (Treatment C), gelcap, orally, once on Day 1 in fasted conditions in Study Period 3. A 14 days washout period was maintained in study period 2 and 3.
  Interventions: Drug: 700 mg resveratrol as JOTROL
- Part 2: JOTROL (Resveratrol) 500 mg (Treatment D) (Experimental): Participants who completed Study Period 3 (Part 1) received JOTROL (resveratrol) 500 (5*100) mg (Treatment D), gelcap, orally, once on Day 1 in fed conditions in Study Period 4. A 14 days washout period was maintained in study period 3 and 4.
  Interventions: Drug: 500 mg resveratrol as JOTROL administered to assess influence of food

INTERVENTIONS:
Drug: 200 mg resveratrol as JOTROL — Low (first) dose of single ascending dose study
  Arms: Part 1: JOTROL (Resveratrol) 200 mg (Treatment A)
Drug: 500 mg resveratrol as JOTROL — Second (intermediate) dose of single ascending dose study
  Arms: Part 1: JOTROL (Resveratrol) 500 mg (Treatment B)
Drug: 700 mg resveratrol as JOTROL — Third (highest) dose of single ascending dose study
  Arms: Part 1: JOTROL (Resveratrol) 700 mg (Treatment C)
Drug: 500 mg resveratrol as JOTROL administered to assess influence of food — 500 mg resveratrol as JOTROL administered to assess influence of food
  Arms: Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)

SUMMARY:
Type of Study: Single Ascending Doses (SAD) Study

Objectives:

To characterize the pharmacokinetic (PK) profile of JOTROL (resveratrol) following oral administration of SAD ranging from 200 mg up to a dose currently estimated at 1,000 mg, in healthy subjects.

To evaluate the safety and tolerability of JOTROL To evaluate the effect of food on the PK profile of JOTROL. Study Design: Phase I, randomized, open-label, sequential SAD study with a food effect evaluation. Blood plasma and urine samples will be assessed for resveratrol and key metabolite content.

Type of Control: No control Test Product: JOTROL (resveratrol) 100 mg resveratrol in 1000 mg softgel capsule for oral administration Dosage Regimen: Planned dose levels of resveratrol: 200 mg, 500 mg, and 1,000 mg. Following completion of each dose level, PK, safety, and tolerability data will be evaluated; dose levels may be adjusted.

Route of Administration: Oral gelcaps with water Number of Subjects: 24 subjects will be included in Part 1; only 16 subjects, who completed Part 1, will be included in Part 2.

Subjects: Healthy, non-smoker, adult males or females, ≥ 18 and ≤ 75 years of age Study Duration: Participation of each subject in this study should last approximately 1 to 1.5 months (for subjects participating in study Part 1 only) and 1.5 to 2 months (for subjects participating in both study parts).

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy male or female volunteers, non-smokers (no use of tobacco products within 3 months prior to screening), ≥ 18 and ≤ 75 years of age, with BMI > 18.5 and < 30.0 kg/m 2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours predose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease as determined by the Investigator.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to study drug administration;
   2. male condom with intravaginally applied spermicide starting at least 21 days prior to study drug administration;
   3. sterile male partner (vasectomized since at least 6 months).
4. Capable of consent

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen or urine cotinine test at screening.
3. History of allergic reactions to resveratrol, polyphenols, other related drugs, .

   or to any excipient in the formulation
4. Positive pregnancy test at screening.
5. Breast-feeding subject.
6. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
7. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
8. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
9. Use of resveratrol for a medical condition or in the context of another clinical trial within a period of 30 days prior to the first dosing.
10. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.

Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

1. prescription medication within 14 days prior to the first dosing;
2. over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 14 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
3. use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration, including St John's wort;
4. depot injection or an implant of any drug within 3 months prior to the first dosing.

12. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.

13. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- inVentiv Health Clinical Research Services LLC, a Syneos Health company (" Syneos Health "), Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kemper C, Benham D, Brothers S, Wahlestedt C, Volmar CH, Bennett D, Hayward M. Safety and pharmacokinetics of a highly bioavailable resveratrol preparation (JOTROL TM). AAPS Open. 2022;8(1):11. doi: 10.1186/s41120-022-00058-1. Epub 2022 Jun 30. PMID 35789594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 21 January 2021 to 31 May 2021.
Pre-assignment Details: A total of 83 healthy participants were screened, of which 29 participants were eligible for this study. Of 29 eligible participants, a total of 24 participants were treated in this single ascending dose study.
Period: Part 1 Study Period 1
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Started | 21 | 0 | 0 | 0
Completed | 16 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Period: Part 1 Study Period 2
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Started | 0 | 16 | 0 | 0
Completed | 0 | 15 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Period: Part 1 Study Period 3
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Started | 0 | 0 | 18 | 0
Completed | 0 | 0 | 15 (3 participants were directly enrolled in Study Period 3 in addition to the 15 participants from the Study Period 2.) | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 2 | 0
Period: Part 2 Study Period 4
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Started | 0 | 0 | 0 | 15
Completed | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all the participants who received at least one dose of the study medication. There were total of 21 participants who started the study as single arm in part 1: Study period 1 and same participants received treatment in the following periods. Only 3 additional participants were enrolled in Part 1, study period 3. Therefore, to avoid double counting of the participants, Baseline data was collected and reported as single arm for all 24 participants.
Groups:
- All Participants: All participants who received JOTROL (resveratrol) 200 (2*100) mg (Treatment A) gelcap, orally once on Day 1 in Study period 1 followed by 500 (5*100) mg (Treatment B) gelcap, orally once on Day 1 in Study period 2 further followed by 700 (7*100) mg (Treatment C) gelcap, orally, on Day 1 in Study period 3 in fasted conditions of Part 1 of the study, followed by JOTROL (resveratrol) 500 (5*100) mg (Treatment D) gelcap, orally, once on Day 1 in fed condition in Study Period 4 of Part 2 of the study. There was a washout period of 14 days between each study period.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence (including clinically significant [CS] vital signs measurements or laboratory results) or worsening of a pre-existing condition in a participant administered a pharmaceutical product during the course of the study, whether related or not to the study medication. TEAEs were defined as AE that occurred on or after the date and time of study drug administration or those that first occurred pre-dose but worsened by increase in occurrence or severity after study drug administration. TEAEs includes both serious and non-serious TEAEs.
Time Frame: From first dose of study drug administration up to 131 days
Population: The safety population was defined as all participants who received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: JOTROL (Resveratrol) 200 mg (Treatment A): Participants received JOTROL (resveratrol) 200 (2*100) mg (Treatment A), gelcap, orally, once on Day 1 in fasted conditions in Study Period 1.
- Part 1: JOTROL (Resveratrol) 500 mg (Treatment B): Participants who completed Study Period 1 received JOTROL (resveratrol) 500 (5*100) mg (Treatment B), gelcap, orally, once on Day 1 in fasted conditions in Study Period 2. A-14 day washout period was maintained in study period 1 and 2.
- Part 1: JOTROL (Resveratrol) 700 mg (Treatment C): Participants who completed Study Period 2 received JOTROL (resveratrol) 700 (7*100) mg (Treatment C), gelcap, orally, once on Day 1 in fasted conditions in Study Period 3. A-14 day washout period was maintained in study period 2 and 3.
- Part 2: JOTROL (Resveratrol) 500 mg (Treatment D): Participants who completed Study Period 3 (Part 1) received JOTROL (resveratrol) 500 (5*100) mg (Treatment D), gelcap, orally, once on Day 1 in fed conditions in Study Period 4. A-14 day washout period was maintained in study period 3 and 4.
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 21 | 16 | 18 | 15
Participants | 7 | 4 | 6 | 6

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Infinity (AUC0-inf) for Resveratrol and Its Metabolites (Resveratrol-3-glucuronide, Resveratrol-4'-Glucuronide, and Resveratrol-3-sulfate)
Description: AUC(0-infinity) of resveratrol, resveratrol-3-glucuronide, resveratrol-4'-glucuronide, and resveratrol-3-sulfate in plasma were reported. AUC(0-infinity) of resveratrol, resveratrol-3-glucuronide, resveratrol-4'-glucuronide, and resveratrol-3-sulfate in plasma were reported and calculated as AUC0-t + Ct/Kel, where Ct is the last observed measurable concentration, AUC0-t is Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration and Kel is Elimination rate constant.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: The pharmacokinetic (PK) population comprised of all participants who received at least one dose of either study drug and had at least one quantifiable PK concentration. "Number analyzed" signifies to participants evaluable for given categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 21 | 16 | 18 | 14
hour*nanogram per milliliter (h*ng/mL)
  Resveratrol: number analyzed (Participants) | 1 | 5 | 3 | 2
  Resveratrol | 214.73 | 499.73 (56.54) | 595.75 (28.19) | 553.77 (60.84)
  Resveratrol-3-Glucuronide | 4821.18 (29.37) | 16390.55 (27.25) | 29570.84 (34.08) | 11834.05 (28.41)
  Resveratrol-3-Sulfate | 11668.98 (27.75) | 35063.90 (31.67) | 53845.25 (20.62) | 31133.94 (33.24)
  Resveratrol-4'-Glucuronide | 4591.06 (27.34) | 15387.06 (29.76) | 22934.42 (29.90) | 14528.02 (21.95)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) for Resveratrol and Its Metabolites (Resveratrol-3-glucuronide, Resveratrol-4'-Glucuronide, and Resveratrol-3-sulfate)
Description: AUC0-t was Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration. AUC(0-t) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: The PK population comprised of all participants who received at least one dose of either study drug and had at least one quantifiable PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 21 | 16 | 18 | 14
h*ng/mL
  Resveratrol | 112.32 (72.49) | 422.85 (53.24) | 785.29 (51.52) | 263.75 (65.72)
  Resveratrol-3-Glucuronide | 4796.08 (29.58) | 16347.62 (27.21) | 29492.22 (34.04) | 11775.27 (28.51)
  Resveratrol-3-Sulfate | 11593.20 (26.78) | 34854.48 (31.49) | 53351.47 (20.04) | 31018.49 (33.26)
  Resveratrol-4'-Glucuronide | 4550.27 (27.58) | 15337.45 (29.70) | 22845.47 (29.36) | 14502.21 (21.93)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Resveratrol and Its Metabolites (Resveratrol-3-glucuronide, Resveratrol-4'-Glucuronide, and Resveratrol-3-sulfate)
Description: Cmax was the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 21 | 16 | 18 | 14
nanogram per milliliter (ng/mL)
  Resveratrol | 94.70 (91.46) | 326.32 (89.76) | 648.08 (73.29) | 140.09 (100.84)
  Resveratrol-3-Glucuronide | 2292.84 (29.69) | 8334.08 (48.84) | 14558.05 (46.33) | 4173.48 (59.28)
  Resveratrol-3-Sulfate | 6204.37 (36.00) | 16863.57 (48.55) | 22856.79 (27.23) | 10696.58 (65.43)
  Resveratrol-4'-Glucuronide | 1649.08 (33.30) | 5340.95 (56.63) | 7663.09 (40.20) | 3742.71 (48.44)

5. Secondary Outcome: Residual Area for Resveratrol
Description: Residual area for resveratrol in plasma was calculated and reported. The residual area was calculated as 100*(1- AUC0-t / AUC0-inf) where AUC0-t (h*ng/mL) = area under the concentration-time curve from time zero to the last measurable concentration and AUC0-inf (h*ng/mL) = area under the plasma concentration-time curve from time 0 to time of infinity.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: PK population comprised of all participants who received at least one dose of either study drug and had at least one quantifiable PK concentration. Here "overall number of participants analyzed" included all participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage AUC
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 1 | 5 | 3 | 2
percentage AUC | 5.48 | 4.56 (73.50) | 3.58 (38.56) | 2.29 (111.16)

6. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Resveratrol
Description: Tmax was time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 21 | 16 | 18 | 14
hour | 0.999 [0.250 to 2.006] | 1.003 [0.496 to 2.001] | 1.025 [0.251 to 2.000] | 1.497 [0.499 to 2.002]

7. Secondary Outcome: Elimination Half-Life (T1/2 el) for Resveratrol
Description: Elimination half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: The PK population comprised of all participants who received at least one dose of either study drug and had at least one quantifiable PK concentration. Here "overall number of participants analyzed" included all participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 1 | 5 | 3 | 2
hour | 1.26 | 2.36 (62.56) | 1.56 (25.19) | 1.47 (71.72)

8. Secondary Outcome: Elimination Rate Constant (Kel) for Resveratrol
Description: Kel was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose and 0.133, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per hour (1/h)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
Number analyzed (Participants) | 1 | 5 | 3 | 2
1 per hour (1/h) | 0.5520 | 0.2932 (48.70) | 0.4436 (28.56) | 0.4712 (71.72)

9. Secondary Outcome: Cumulative Urinary Excretion From Time Zero to Time t (Ae0-t) for Resveratrol
Description: Cumulative urinary excretion from time zero to time t, calculated as the sum of the amounts excreted over each collection interval. The amount excreted in urine for each time interval was calculated as the urine concentration multiplied by the urine volume.
Time Frame: Pre-dose and 4, 8, 12, 24, and 32 hours post-dose on Day 1
Population: The PK population comprised of all participants who received at least one dose of either study drug and had at least one quantifiable PK concentration. As pre-specified, this outcome measure was planned to be assessed for Part 1 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C)
Number analyzed (Participants) | 21 | 16 | 18
nanogram (ng) | 16927.35 (75.39) | 48454.76 (49.88) | 109323.50 (88.32)

10. Secondary Outcome: Maximum Rate of Urinary Excretion (Rmax) for Resveratrol
Description: Maximum rate of urinary excretion, calculated by dividing the amount of drug excreted in each collection interval by the time over which it was collected.
Time Frame: Pre-dose and 4, 8, 12, 24, and 32 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per hour (ng/h)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C)
Number analyzed (Participants) | 21 | 16 | 18
nanogram per hour (ng/h) | 8791.49 (82.45) | 26486.23 (136.58) | 44737.57 (90.97)

11. Secondary Outcome: Time of Rmax (Tmax) for Resveratrol
Description: Tmax was the time after administration of a drug when the Rmax is reached.
Time Frame: Pre-dose and 4, 8, 12, 24, and 32 hours post-dose on Day 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C)
Number analyzed (Participants) | 21 | 16 | 18
hour | 0.793 [0.233 to 12.013] | 0.551 [0.049 to 1.436] | 0.698 [0.290 to 3.563]

12. Secondary Outcome: Renal Clearance (CLr) for Resveratrol
Description: CLr was calculated as Ae0-t/AUC0-t (plasma) where t is Tlast.
Time Frame: Pre-dose and 4, 8, 12, 24, and 32 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C)
Number analyzed (Participants) | 21 | 16 | 18
liter per hour (L/h) | 0.15 (112.22) | 0.11 (63.04) | 0.14 (95.39)

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to 131 days
Arm/Group | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/16 | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/16 | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 7/21 | 4/16 | 6/18 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: JOTROL (Resveratrol) 200 mg (Treatment A) (N=21) | Part 1: JOTROL (Resveratrol) 500 mg (Treatment B) (N=16) | Part 1: JOTROL (Resveratrol) 700 mg (Treatment C) (N=18) | Part 2: JOTROL (Resveratrol) 500 mg (Treatment D) (N=15)
Somnolence (Nervous system disorders) | 3 | 2 | 2 | 2
Headache (Nervous system disorders) | 3 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0
White blood cells urine (Investigations) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04668274/Prot_003.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT04668274/SAP_004.pdf
  • Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04668274/ICF_002.pdf